CLINICAL TRIAL: NCT01412827
Title: Diagnostic and Prognostic Accuracy of Stress SPECT Myocardial Perfusion Imaging With Half the Usual Radiotracer Dose
Brief Title: Accuracy of Half of the Usual Radiotracer Dose in SPECT
Acronym: SPECT-Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Renee Hessian, Dr. Renee Hessian, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HI Protocol #2010127-01H
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
Keywords: Single-photon emission computed tomography; myocardial perfusion imaging; rest/stress; treadmill; persantine; half-dose; radiotracer; tetrofosmin; Thallium; cadmium zinc telluride; diagnostic; prognostic
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Comparison of radioisotope dosing (Other)
  Interventions: Radiation: 1/2 dose of 99mTc OR 201Tl tracers

INTERVENTIONS:
Radiation: 1/2 dose of 99mTc OR 201Tl tracers — Rest: Imaging will occur 30 to 60 minutes after injection of tracer.
  Stress: All patients will undergo a symptom-limited Bruce protocol treadmill exercise test. At peak stress, the radiotracer will be injected intravenously, and exercise will continue for an additional 60 s. The patients who are unable to achieve the targeted heart rate or exercise will be stressed pharmacologically. Dipyridamole (0.142 mg/kg/min) will be infused intravenously for 5 minutes, and 99mTc radiotracer will be injected at 2 min after infusion completion (7 min into the study). Aminophylline (100-200 mg) will be given intravenously 2 min after injection of the radiotracer.

SUMMARY:
There has been a shortage of nuclear isotopes, not only in Canada but around the world. New, more sensitive SPECT cameras can obtain better images in shorter scan times. These cameras have also shown the ability to use a smaller dose of radioisotope to obtain the images. New software has been tested on the standard camera, the GE Infinia-Hawkeye SPECT/CT. The Diagnostic Imaging Department of The University of Ottawa Heart Institute has also acquired a new camera, the Discovery NM530c CZT and has been doing heart scans in shorter times. The investigators will now be looking at the quality of images using less isotope during SPECT myocardial perfusion imaging for diagnostic and prognostic purposes.

DETAILED DESCRIPTION:
SPECT MPI is well accepted as a reliable and cost-effective tool for diagnosis, risk stratification and management of patients with suspected or known coronary artery disease (CAD) (1;2). MPI represents approximately 40% of nuclear medicine patient studies and most of these use 99mTc-sestamibi or 99mTc-tetrofosmin(3). Rest/stress MPI using 99mTc-sestamibi and 99mTc-tetrofosmin uses more tracer doses than many other nuclear medicine tests and thus account for >50% of injected radiotracer activity(3). Thus, interruptions in the supply of 99Mo, the parent isotope of 99mTc, significantly affect stress MPI imaging and associated patient care.

Alternatives to 99mTc-sestamibi and 99mTc-tetrofosmin for perfusion imaging include 201Tl for SPECT imaging and 82Rb or 13NH3 for positron emission tomography (PET) imaging (4;5). MPI using 201Tl has similar diagnostic accuracy but image interpretation is more difficult due to greater scatter and attenuation. Moreover, the patient effective radiation dose for MPI using a standard injected dose of 3.5mCi of 201Tl is ~20 mSv. This radiation dose is twice that of 99mTc tracers which typically deliver an effective dose of ~10 mSv. PET imaging with 82Rb or 13NH3 is another alternative, but is much more expensive and not routinely available in Canada due to a very limited install base of PET scanners and associated cyclotrons. The number of SPECT cameras operational in Canada is more than 40 times the number of PET scanners.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting for clinically indicated SPECT perfusion scan
* Patients presenting to sites with a functional CZT camera. Available sites are Ottawa (OHI), Mississauga, and Calgary.
* Age >18 years old

Exclusion Criteria:

* Patients with a life expectancy less than 1 year, from non cardiac cause
* Age < 18 years old or lack of consent
* Allergy or contraindication to dipyridamole
* Refractory angina or infarction or need for urgent angiography
* Known pregnancy
* Uncontrolled atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of non-fatal infarction or death in the normal group of SPECT-Light acquisitions versus standard SPECT acquisitions | 2 years
  The difference in the rate of non-fatal infarction or death that occurs in the normal group of the combined SPECT-Light acquisition protocols (LDa and LDb) versus the outcome that occurs in the acquisitions obtained by the standard SPECT (FD) protocol.

SECONDARY OUTCOMES:
Comparison of classification of the degree of abnormality based on the two image acquisition protocols | 2 years
  A comparison of classification of the degree of abnormality based on the two image acquisition protocols. Multi-level correlation between the two image sets (LDa vs 2 and LDb vs 2) will be obtained against the standard SPECT (FD) images.
  The combined rates of non-fatal MI or death in each of the LD images as well as the standard dose images (FD) which are considered abnormal (SSS ≥ 4) will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Renée Hessian, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Hachamovitch R, Hayes SW, Friedman JD, Cohen I, Berman DS. Stress myocardial perfusion single-photon emission computed tomography is clinically effective and cost effective in risk stratification of patients with a high likelihood of coronary artery disease (CAD) but no known CAD. J Am Coll Cardiol. 2004 Jan 21;43(2):200-8. doi: 10.1016/j.jacc.2003.07.043. PMID 14736438
- [Background] Marcassa C, Bax JJ, Bengel F, Hesse B, Petersen CL, Reyes E, Underwood R; European Council of Nuclear Cardiology (ECNC); European Society of Cardiology Working Group 5 (Nuclear Cardiology and Cardiac CT); European Association of Nuclear Medicine Cardiovascular Committee. Clinical value, cost-effectiveness, and safety of myocardial perfusion scintigraphy: a position statement. Eur Heart J. 2008 Feb;29(4):557-63. doi: 10.1093/eurheartj/ehm607. Epub 2008 Jan 17. PMID 18202253
- [Background] Beanlands RS, Chow BJ, Dick A, Friedrich MG, Gulenchyn KY, Kiess M, Leong-Poi H, Miller RM, Nichol G, Freeman M, Bogaty P, Honos G, Hudon G, Wisenberg G, Van Berkom J, Williams K, Yoshinaga K, Graham J; Canadian Cardiovascular Society; Canadian Association of Radiologists; Canadian Association of Nuclear Medicine; Canadian Nuclear Cardiology Society; Canadian Society of Cardiac Magnetic Resonance. CCS/CAR/CANM/CNCS/CanSCMR joint position statement on advanced noninvasive cardiac imaging using positron emission tomography, magnetic resonance imaging and multidetector computed tomographic angiography in the diagnosis and evaluation of ischemic heart disease--executive summary. Can J Cardiol. 2007 Feb;23(2):107-19. doi: 10.1016/s0828-282x(07)70730-4. PMID 17311116